CLINICAL TRIAL: NCT05011175
Title: Exercise Habits: A Survey of Individuals With Parkinson's Disease Living in the Community
Status: Completed | Type: Observational
Sponsor: Jordana Lockwich (Other)
Responsible Party: Sponsor-Investigator, Jordana Lockwich, Graduate Student, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 59258
Record Dates: First submitted 2021-08-16; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: Exercise; Survey
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Parkinson's Disease: Individuals that have been diagnosed with Parkinson's Disease will be enrolled to participant in the survey research.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Participants responded to questions about their exercise habits and perceived levels of intensity as well as demographic information.

SUMMARY:
This study aims to evaluate the exercise regimens of individuals with Parkinson's.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's Disease
* Able to speak English

Exclusion Criteria:

* No internet access

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals ages 40-90 years old who have been diagnosed with Parkinson's Disease.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Age | Reported at baseline
  Average age of participants enrolled
Self-reported age of Parkinson's Disease Diagnosis | Reported at baseline
  Average age of diagnosis with Parkinson's Disease for enrolled participants.
Self-reported education level | Reported at baseline
  Number of participants reporting 1. less than 12 years of school, 2. completed high school, 3. completed bachelor degree, 4. completed graduate/advanced degree.
Self-reported living situation | Reported at baseline
  Number of participants reporting 1.living alone, 2. living with others 3. living in a healthcare facility
Self-reported number of years taking medicine for Parkinson's Disease | Reported at baseline
  Average number of years participants reported taking medication for Parkinson's Disease
Self-reported brain stimulation treatment | Reported at baseline
  Number of participants reporting they have undergone deep brain stimulation for Parkinson's Disease.
Self-reported stage of Parkinson's Disease | Reported at baseline
  Average reported stage of Parkinson's Disease participants (1. mild with no symptoms, 2. mild with symptoms, 3. moderate, 4. advanced, able to walk 5. advanced, unable to walk).
Self-reported physical help requirement | Reported at baseline
  Number of participants reporting 1. they need help from another person during the day or 2. they do not need help from another person during the day.
Self-reported walking ability | Reported at baseline
  Number of participants reporting 1. ability to walk unaided, 2. ability to walk with an assistive device, or 3. requiring assistance to walk
Self-reported mobility level | Reported at baseline
  Participants reported mobility level ranging from independent to total assist required.
Self-reported current exercise habits survey | Reported at baseline
  3 question survey component evaluating the exercise habits of individuals with Parkinson's Disease using a Likert scale from 0-5 where 5 indicated a higher levels of exercise.
Perceived levels of intensity | Reported at baseline
  7 question survey evaluating the level of intensity of exercise of individuals with Parkinson's Disease using a Likert scale from 0-5 where 5 indicated higher levels of intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Lockwich, PT, DPT, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No